CLINICAL TRIAL: NCT01188798
Title: Methotrexate or Pentostatin for Graft-versus-host Disease Prophylaxis in Risk-adapted Allogeneic Bone Marrow Transplantation for Hematologic Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUDSIB
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2012-02

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelocytic Leukemia; Chronic Myelocytic Leukemia; Hodgkin's Disease; Myelodysplastic Syndrome
Keywords: Allogeneic Bone Marrow Transplantation; Graft versus host disease; Tacrolimus; Sirolimus; Methotrexate; Pentostatin
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease; Myelodysplastic Syndromes; Graft vs Host Disease | interventions — Methotrexate; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transplant recipients receiving Methotrexate (Experimental): Participants will be biologically stratified according to disease, donor, and KIR match. In addition to a standard backbone of 2 GVHD prophylactics, a computer generated randomization procedure will assign participants to a third GVHD prophylactic medication (MTX or pentostatin)
  Interventions: Drug: Methotrexate
- Transplant recipients receiving Pentostatin (Experimental): Participants will be biologically stratified according to disease, donor, and KIR match.between donor and host.In addition to a standard backbone of 2 GVHD prophylactics, a computer generated randomization procedure will assign participants to a third GVHD prophylactic medication (MTX or pentostatin)
  Interventions: Drug: Pentostatin

INTERVENTIONS:
Drug: Methotrexate — Participants will be randomized to receive either methotrexate (MTX) or pentostatin for graft-versus-host disease (GVHD) prophylaxis after receiving an allogeneic bone marrow transplant from an HLA-matched related or unrelated donor.
  Arms: Transplant recipients receiving Methotrexate
Drug: Pentostatin — Participants will be randomized to receive either methotrexate (MTX) or pentostatin for graft-versus-host disease (GVHD) prophylaxis after receiving an allogeneic bone marrow transplant from an HLA-matched related or unrelated donor.
  Arms: Transplant recipients receiving Pentostatin

SUMMARY:
The purpose of the study is to determine if participants who receive the GVHD prophylaxis medication pentostatin will have less severe hepatic toxicities than those receiving MTX. The study is estimated to have sufficient statistical power to ascertain at least a 20% improvement in day 42 NCI CTC grade 2 or above hepatic toxicity-free survival in pentostatin recipients.

DETAILED DESCRIPTION:
Participants will be randomized to receive either methotrexate (MTX) or pentostatin for graft-versus-host disease (GVHD) prophylaxis after receiving an allogeneic bone marrow transplant from an HLA-matched related or unrelated donor. All participants will receive a standard backbone GVHD prophylaxis regimen (tacrolimus and sirolimus) and conditioning (cyclophosphamide/TBI). A risk-adapted approach will be used during conditioning to further minimize the risk of leukemia relapse based on two factors:

1. Lymphoid versus myeloid primary disease.
2. KIR compatibility between donor and host.

ELIGIBILITY:
Inclusion Criteria:

*Age less than or equal to 21 years old

High risk malignancy as follows:

* High-risk ALL in CR1. Examples include, but not limited to: Induction failure or > 1% leukemic lymphoblasts in the bone marrow on remission date;> 0.1% leukemic lymphoblasts in the bone marrow in week 7 of continuation treatment (i.e. before reinduction I); re-emergence of leukemic lymphoblasts by MRD (at any level) in patients previously MRD negative; persistently detectable MRD at lower levels;early T-cell precursor (ETP) ALL.
* High-risk ALL beyond CR1, or with refractory disease. "Beyond CR1" denotes any CR following CR1, or any relapsed state. "Refractory disease" includes induction failure.
* High-risk de novo AML in CR1.Examples include but are not limited to:evidence of a high-risk genetic abnormality or high-risk MRD features.
* AML beyond CR1, or with refractory disease. "Beyond CR1" denotes any CR following CR1, or any relapsed state. "Refractory disease" includes induction failure.
* Therapy-related AML.
* MDS, primary or secondary, at any stage.
* NK cell lymphoblastic leukemia in any CR
* Biphenotypic bilineage, or undifferentiated leukemia.
* CML in any phase
* Hodgkin lymphoma beyond CR1 or with refractory disease. "Beyond CR1" denotes any CR following CR1, or any relapsed state.
* Non-Hodgkin lymphoma beyond CR1 or with refractory disease. "Beyond CR1" denotes any CR following CR1, or any relapsed state.
* Juvenile Myelomonocytic Leukemia (JMML).
* All patients with prior evidence of CNS leukemia must be treated and be in CNS CR to be eligible for study.
* Has a suitable HLA matched sibling or unrelated volunteer donor available for stem cell donation.A "matched" donor is defined as allele matching at 7/8 to 8/8 HLA loci at A, B, C and DRB1.For the purpose of this study, the term "matched sibling" also refers to an HLA matched family member.
* Does not have any other active malignancy other than the one for which this transplant is indicated.
* Left ventricular ejection fraction > 40%,or shortening fraction > 26%.
* Forced vital capacity (FVC) greater than or equal to 50% of predicted value (corrected for hemoglobin), or if patient is unable to perform pulmonary function testing, pulse oximetry greater than or equal to 92% on room air.
* Creatinine clearance greater than or equal to 70 ml/min/1.73m2
* Karnofsky or Lansky (age-dependent) performance score of greater than or equal to 70.
* Bilirubin less than or equal to 2.5 mg/dL.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than or equal to 5 times upper limit of normal
* Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment.
* Not lactating.
* Has not had a prior allogeneic HSCT.

Exclusion Criteria:

* Pregnant and lactating females are excluded from participation as the short and long-term effects of the protocol interventions and infusion on a fetus or a nursing child through breast milk are not entirely known at this time.

Ages: 18 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asha Pillai, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six transplant patients were recruited between December, 2010 through March, 2011. Participants will be biologically stratified according to disease, donor, and KIR match.
Groups:
- Methotrexate: Participants will be biologically stratified according to disease, donor, and KIR match. In addition to a standard backbone of 2 GVHD prophylactics, a computer generated randomization procedure will assign participants to a third GVHD prophylactic medication (MTX or pentostatin)
  Participants were randomized to receive methotrexate (MTX) for graft-versus-host disease (GVHD) prophylaxis after receiving an allogeneic bone marrow transplant from an HLA-matched related or unrelated donor.
- Pentostatin: Participants will be biologically stratified according to disease, donor, and KIR match between donor and host. In addition to a standard backbone of 2 GVHD prophylactics, a computer generated randomization procedure will assign participants to a third GVHD prophylactic medication (MTX or pentostatin)
  Participants were randomized to receive pentostatin for graft-versus-host disease (GVHD) prophylaxis after receiving an allogeneic bone marrow transplant from an HLA-matched related or unrelated donor.
Period: Overall Study
Arm/Group | Methotrexate | Pentostatin
Started | 2 | 4
Completed | 0 | 1
Not Completed | 2 | 3
Not completed — Death | 0 | 1
Not completed — Required additional transplant | 1 | 1
Not completed — Protocol closure | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Methotrexate: Participants will be biologically stratified according to disease, donor, and KIR match. In addition to a standard backbone of 2 GVHD prophylactics, a computer generated randomization procedure will assign participants to a third GVHD prophylactic medication (MTX or pentostatin)
  Methotrexate: Participants were randomized to receive methotrexate (MTX) for graft-versus-host disease (GVHD) prophylaxis after receiving an allogeneic bone marrow transplant from an HLA-matched related or unrelated donor.
- Pentostatin: Participants will be biologically stratified according to disease, donor, and KIR match between donor and host. In addition to a standard backbone of 2 GVHD prophylactics, a computer generated randomization procedure will assign participants to a third GVHD prophylactic medication (MTX or pentostatin)
  Pentostatin: Participants were randomized to receive pentostatin for graft-versus-host disease (GVHD) prophylaxis after receiving an allogeneic bone marrow transplant from an HLA-matched related or unrelated donor.
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Pentostatin | Total
Number analyzed (Participants) | 2 | 4 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 10.35 (0.07) | 12.95 (6.65) | 12.08 (5.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Determining Whether the Hepatic Adverse Event-free (NCI Grades II-IV) Survival at Day 42 After an HLA-matched Transplant for Hematologic Malignancy Can be Improved by Using a GVHD Prophylaxis Regimen That Includes Pentostatin Rather Than MTX.
Description: The hypothesis was that individuals receiving the drug pentostatin as GVHD prophylaxis would experience less severe hepatic toxicity than those receiving methotrexate as GVHD prophylaxis. The study is estimated to have sufficient statistical power to ascertain at least a 20% improvement in day 42 grade 2 or above hepatic toxicity-free survival in pentostatin recipients
Time Frame: 42 days post-transplant
Population: Insufficient data was available to answer objectives
Groups:
- Methotrexate: Participants will be biologically stratified according to disease, donor, and KIR match. In addition to a standard backbone of 2 GVHD prophylactics, a computer generated randomization procedure will assign participants to a third GVHD prophylactic medication (MTX or pentostatin)
  Merthotrexate: Participants were randomized to receive methotrexate (MTX) for graft-versus-host disease (GVHD) prophylaxis after receiving an allogeneic bone marrow transplant from an HLA-matched related or unrelated donor.
Arm/Group | Methotrexate | Pentostatin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Assess Overall Survival, Relapse, Engraftment, and Regimen-related Morbidity and Estimating Cumulative Incidence of Pulmonary Adverse Events and Mucositis.
Description: To characterize the pharmacokinetic-pharmacodynamic relationships of pentostatin in this patient population and to assess the relationship between pre-transplant minimal residual disease (MRD) and transplant outcomes.
Time Frame: 42 days post- transplant
Population: Insufficient data was available to answer objectives.
Groups:
- Pentostatin: Participants will be biologically stratified according to disease, donor, and KIR match between donor and host. In addition to a standard backbone of 2 GVHD prophylactics, a computer generated randomization procedure will assign participants to a third GVHD prophylactic medication (MTX or pentostatin).
  Pentostatin: Participants were randomized to receive pentostatin for graft-versus-host disease (GVHD) prophylaxis after receiving an allogeneic bone marrow transplant from an HLA-matched related or unrelated donor.
Arm/Group | Methotrexate | Pentostatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from diagnosis to day 100 post-transplant.
Arm/Group | Methotrexate | Pentostatin
Serious Adverse Events (participants affected / at risk) | 2/2 | 4/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate (N=2) | Pentostatin (N=4)
Graft Versus Host Disease (GVHD), Acute, Liver (Immune system disorders) | 0 (0) | 1 (1)
Graft Versus Host Disease (GVHD), Joint, Chronic (Immune system disorders) | 0 (0) | 1 (1)
Fever without Neutropenia (General disorders) | 2 (4) | 2 (3)
Ulcer of pharynx (disorder) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Failure, Hepatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Veno-occlusive Disease, Hepatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Infection, Klebsiella, Blood (Infections and infestations) | 0 (0) | 1 (1)
Anemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Encephalopathy due to vitamin deficiency (disorder) (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate (N=2) | Pentostatin (N=4)
Cytokine Release Syndrome (Stem Cell Infusion) (Immune system disorders) | 0 (0) | 2 (2)
Cytokine Release Syndrome (Thymoglobulin) (Immune system disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Fever without Neutropenia (General disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chronic gastritis (disorder) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gallbladder Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (finding) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulcer of pharynx (disorder) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (disorder) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bleeding/Hemorrhage, Gastrointestinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Hematemesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhagic Cystitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Typhlitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 2 (5) | 1 (1)
Infection, Adenovirus, Blood (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infection, Adenovirus, Stool (Infections and infestations) | 1 (1) | 1 (1)
Infection, BK Virus, Blood (Infections and infestations) | 0 (0) | 2 (2)
Infection, BK Virus, Urine (Infections and infestations) | 0 (0) | 1 (1)
Infection, Clostridium Difficile, Stool (Infections and infestations) | 2 (2) | 1 (1)
Infection, Cytomegalovirus, Urine (Infections and infestations) | 0 (0) | 1 (1)
Infection, E. Coli, Blood (Infections and infestations) | 0 (0) | 1 (1)
Infection, Helicobacter pylori, Stomach (Infections and infestations) | 1 (1) | 0 (0)
Infection, Herpes Simplex Virus (HSV), Oral (Infections and infestations) | 0 (0) | 1 (1)
Infection, Pseudomonas Aeruginosa, Blood (Infections and infestations) | 0 (0) | 1 (1)
Infection, Staphylococcus Epidermidis, Blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, Varicella Zoster, Abdomen, Skin (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Hypertension (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic Encephalopathy (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mood Alteration (Nervous system disorders) | 1 (1) | 0 (0)
Sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nodule, Pulmonary, Left Lower Lobe (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Disease, Renal (Renal and urinary disorders) | 0 (0) | 1 (1)
Engraftment Syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated prematurely. The Data Safety and Monitoring Board (DSMB) requested major scientific study changes. This was deemed infeasible by institutional leadership and study was terminated. Therefore, no final results exist to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes